CLINICAL TRIAL: NCT03759132
Title: Effects of Transcranial Direct Current Stimulation on Postural Control: a Double-blind Randomized Controlled Trial.
Brief Title: Effects of Transcranial Direct Current Stimulation on Postural Control
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS in Parkinson's Disease
Record Dates: First submitted 2018-11-21; First posted 2018-11-29 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): Bihemispheric tDCS applied over primary motor cortex.
  Dose: 2mA, 20 minutes
  Interventions: Procedure: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Bihemispheric tDCS applied over primary motor cortex.
  Dose: 2mA, 20 minutes (30s ON)
  Interventions: Procedure: Transcranial direct current stimulation

INTERVENTIONS:
Procedure: Transcranial direct current stimulation — Transcranial direct current stimulation is a noninvasive technique of neuronal modulation that has been used in different chronic neurological conditions, including Parkinson's disease.

SUMMARY:
Parkinson's disease is a progressive, degenerative neurological disease associated with profound changes in the quality of life of its survivors. Recent evidence has demonstrated the potential use of transcranial direct current stimulation (tDCS) to modulate cerebral excitability and movement control in neurological chronic conditions. However, few studies have investigated the effects of tDCS on postural control in patients with Parkinson's disease. This study aims to investigate the effect of bihemispheric tDCS on postural control in people with Parkinson's disease. Participants will be randomized to receive a single session of anodal and sham bihemispheric tDCS (7 days between each type of stimulation).

Primary clinical outcome (balance) will be collected before and immediately after tDCS. The data will be collected by a blind examiner to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

Medical diagnosis of idiopathic Parkinson's disease present for at least 12 months

In clinical follow-up and pharmacological treatment by a responsible physician

Parkinson's classification of 1.5-3 according to the Hoehn and Yahr scale

Signing of the free and informed consent form-

Exclusion Criteria:

Use any associated orthopedic device to aid gait or balance control

Signs of severe dementia (evaluated by the Mini-Mental State Examination - MMSE)

Diagnosis of other neurological disorders (including those of central and peripheral nature)

Previous treatment with tDCS

Medical diagnosis of psychiatric illnesses with the use of centrally acting medications (depressants)

The use of pacemakers or other implanted devices.-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change from COP - AP axis | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) in antero-posterior (AP) axis in centimeters.
Change from COP - ML axis | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) in Mediolateral (ML) axis in centimeters.
Change from COP - area | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) area (cm²).

OTHER OUTCOMES:
Adverse effects | Immediately after tDCS
  Adverse effects will be evaluated using structured questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No